CLINICAL TRIAL: NCT03594890
Title: A First-in-human Phase I, Single Center, Randomized, Observer-blind, Placebo-controlled Study to Evaluate the Safety and Immune Response of Increasing Doses of OVX836 Vaccine After Intramuscular (IM) or Intranasal (IN) Administrations in Healthy Subjects Aged 18-49 Years.
Brief Title: Safety and Immune Response of Increasing Doses of OVX836 After Intramuscular or Intranasal Administrations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Osivax (Industry)
Collaborators: Aepodia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: OVX836-001
Record Dates: First submitted 2018-06-20; First posted 2018-07-20 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Influenza
Keywords: influenza; vaccine; nucleoprotein
MeSH Terms: conditions — Influenza, Human | interventions — Injections, Intramuscular

STUDY DESIGN:
Intervention Model Description: Phase I, single center, randomized, observer-blind, placebo-controlled study.
Who Masked: Participant, Investigator
Masking Description: This study will be an observer-blind study with the subject-blind and the investigator-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OVX836 (Intramuscular) (Experimental): OVX836 is a recombinant Influenza vaccine based on the NP of the Influenza virus. OVX836 vaccine is a ready to use sterile liquid clear and colourless solution, presented in 2 mL glass vials filled with 1.2 mL solution. It contains 300 µg/mL of OVX836 vaccine and is formulated without adjuvant.
  3 Dose levels tested: 30µg, 90 µg and 180 µg.
  Interventions: Biological: OVX836 (Intramuscular)
- Placebo (Intramuscular) (Placebo Comparator): The Placebo, is Sodium Chloride 0.9 % ready to use sterile solution. The volume of placebo to be administered will be similar to the one of the experimental vaccine.
  Interventions: Biological: Placebo (Intramuscular)
- OVX836 (Intranasal) (Experimental): OVX836 is a recombinant Influenza vaccine based on the NP of the Influenza virus. OVX836 vaccine is a ready to use sterile liquid clear and colourless solution, presented in 2 mL glass vials filled with 1.2 mL solution. It contains 300 µg/mL of OVX836 vaccine and is formulated without adjuvant.
  3 Dose levels tested: 30µg, 90 µg and 180 µg.
  Interventions: Biological: OVX836 (Intranasal)
- Placebo (Intranasal) (Placebo Comparator): The Placebo, is Sodium Chloride 0.9 % ready to use sterile solution. The volume of placebo to be administered will be similar to the one of the experimental vaccine.
  Interventions: Biological: Placebo (Intranasal)

INTERVENTIONS:
Biological: OVX836 (Intramuscular) — 2 consecutive administrations of OVX836 vaccine at Day 1 and Day 29.
  Arms: OVX836 (Intramuscular)
Biological: Placebo (Intramuscular) — 2 consecutive administrations of placebo at Day 1 and Day 29.
  Arms: Placebo (Intramuscular)
Biological: OVX836 (Intranasal) — 2 consecutive administrations of OVX836 vaccine at Day 1 and Day 29.
  Arms: OVX836 (Intranasal)
Biological: Placebo (Intranasal) — 2 consecutive administrations of placebo at Day 1 and Day 29.
  Arms: Placebo (Intranasal)

SUMMARY:
The present study is a first-in-man clinical trial evaluating OVX836, a recombinant broad spectrum vaccine for Influenza.

This clinical trial will evaluate the safety and the immune response of increasing doses of OVX836 after intramuscular or intranasal administrations in healthy volunteers.

DETAILED DESCRIPTION:
This study is a single center, randomized, sequential dose escalation, placebo-controlled, observer-blind study conducted in healthy subjects aged 18-49 years.

The OVX836 recombinant vaccine is based on the well conserved nucleoprotein of the Influenza virus.

Three different dose levels of OVX836 (30µg, 90µg, 180µg) will be assessed sequentially and administered either by the intramuscular route (Study Part A) or by the intranasal route (Study Part B).

There will be 6 cohorts in total with one cohort testing one dose level and one route of administration. Each study cohort will be composed of 12 subjects, with 9 subjects receiving the OVX836 vaccine and 3 subjects receiving the placebo. Each subject will receive one administration of OVX836 or placebo on Day 1 and one administration on Day 29.

The study duration for each subject is approximately 5 months.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent approved by the relevant Ethical Committee governing the site.
2. Overtly healthy male or female subjects, as determined by medical history and medical examination.
3. Between the ages of 18 and 49 years, inclusive, on screening.
4. Between the Body Mass Index of 18 and 24 kg/m2, inclusive, on screening.
5. Clinical laboratory test results within normal reference range, or results with acceptable deviations that are judged to be Non Clinically Significant by the Investigator.
6. Blood Pressure and Heart Rate within normal reference range, or results with acceptable deviations that are judged to be Non Clinically Significant by the Investigator.
7. Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.

Exclusion Criteria:

1. Previous Influenza vaccination within the 6 months before screening.
2. History of significant medical illness such as auto immune diseases, immune deficiency, uncontrolled diabetes or hypertension, heart or renal or hepatic diseases, as judged by the investigator.
3. For female subjects: pregnant or breast-feeding or of childbearing potential without appropriate contraceptive methods or with positive pregnancy test at screening.
4. Having received another vaccination within 3 months prior to screening.
5. Plan to receive other vaccine during the study period.
6. Administration of any investigational or non-registered drug or vaccine within 3 months prior to the first administration of study vaccine.
7. History of receiving blood or blood component or IgG within 3 months prior to screening.
8. Presence of acute febrile illness (temperature > 38°C, temporary exclusion criteria).
9. For intranasal route: common cold and rhinitis (temporary exclusion criteria).
10. Individuals with any progressive or severe neurological disorder, seizure disorder or Guillain-Barré syndrome.
11. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the Investigator, may interfere with the subject's ability to participate in the study.
12. History of alcoholism and/or drug abuse or tabagism (above 10 cigarettes a day).
13. Treatment that can affect immune response such as systemic or high dose inhaled corticosteroids (>800µg/day beclometasone or equivalent), radiation treatment, cytotoxic drugs or chronic non-steroidal anti-inflammatory drugs (more than 4 weeks), interferon, immunomodulators, allergy shots, as judged by the Investigator.
14. Positive test for HIV, HBV or HCV at screening.
15. History of severe allergic reactions and/or anaphylaxis or serious adverse reactions to vaccines and antibiotics.
16. Any contraindication to intranasal or intramuscular administration, as judged by the Investigator.
17. Individuals with history of any illness that, in the opinion of the Investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
18. Sponsor employees or Investigator site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Out-of-Range Safety Lab data | 28 days after last vaccine administration.
  Frequency (number and percentage) of subjects with deviations from normal values of hematological and biochemical blood tests
Safety: Solicited local and systemic reactions | 7 days after last vaccine administration.
  Frequency (number and percentage) of subjects with reported solicited local and systemic reactions
Safety: Unsolicited Adverse Events | 28 days after last vaccine administration.
  Frequency (number and percentage) of subjects with reported unsolicited Adverse Event (AE)
Safety: Serious Adverse Events | at end of study visit (i.e. Week 22)
  Frequency (number and percentage) of subjects with reported Serious Adverse Event (SAE)

SECONDARY OUTCOMES:
Immune response: frequency of subjects with anti-NP IgG antibody titres | 28 days post each vaccine administration and 5 months after the 1st vaccine administration (i.e. Day 29, Day 57, Day 150) versus Day 1 pre-dose.
  Frequency (number and percentage) of subjects with an increase of anti-NP Immunoglobulin G (IgG) (ELISA, serum) for each dose level of OVX836 administered by the intramuscular or intranasal route.
Immune response: anti-NP IgG antibody titres (geometric mean) | 28 days post each vaccine administration and 5 months after the 1st vaccine administration (i.e. Day 29, Day 57, Day 150) versus Day 1 pre-dose.
  Geometric Mean in anti-NP Immunoglobulin G (IgG) (ELISA, serum) for each dose level of OVX836 administered by the intramuscular or intranasal route.
Immune response: frequency of subjects with anti-NP IgA antibody titres | 28 days post each vaccine administration and 5 months post 1st vaccine administration (e.g. Day 29, Day 57, Day 150) versus Day 1 pre-dose.
  Frequency (number and percentage) of subjects with an increase of Anti-NP Immunoglobulin A (IgA) (ELISA, nasal swab) for each dose level of OVX836 administered by the intranasal route.
Immune response: anti-NP IgA antibody titres (geometric mean) | 28 days post each vaccine administration and 5 months post 1st vaccine administration (e.g. Day 29, Day 57, Day 150) versus Day 1 pre-dose.
  Geometric Mean in anti-NP Immunoglobulin A (IgA) (ELISA, serum) for each dose level of OVX836 administered by the intranasal route.
Immune response: frequency of subjects with NP T cell resoonse | Day 1 pre-dose, 7 days and 28 days post each vaccine administration, and 5 months post 1st vaccine administration (e.g. Day 1, Day 8, Day 29, Day 36, Day 57, Day 150).
  Frequency (number and percentage) of subjects with NP T cell response (ELISPOT, Peripheral Blood Mononuclear Cells (PBMC)) for each dose level of OVX836 by the intramuscular or intranasal route.
Immune response: mean NP T cell response | Day 1 pre-dose, 7 days and 28 days post each vaccine administration, and 5 months post 1st vaccine administration (e.g. Day 1, Day 8, Day 29, Day 36, Day 57, Day 150).
  NP T cell response (mean ELISPOT counts) for each dose level of OVX836 administered by the intramuscular or intranasal route.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, MD, PhD, Principal Investigator — Centre for the Evaluation of Vaccination, University of Antwerp
Locations (1):
- Centre for the Evaluation of Vaccination, University of Antwerp, Antwerp, Belgium

REFERENCES:
- See also: Sponsor — http://www.osivax.com/
- See also: Clinical Unit — https://www.uantwerpen.be/en/research-groups/vaxinfectio/
- See also: Phase 1 Randomized, Placebo-Controlled, Dose-Escalating Study to Evaluate OVX836, a Nucleoprotein-Based Influenza Vaccine: Intramuscular Results — https://pubmed.ncbi.nlm.nih.gov/34653245/